CLINICAL TRIAL: NCT06759948
Title: An Early Exploratory Clinical Study of GC012F Injection in the Treatment of Refractory Generalized Myasthenia Gravis
Acronym: KY2024-853
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongbo Zhao (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chongbo Zhao, Chief Physician of Neurology, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-853
Record Dates: First submitted 2024-12-19; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Generalized Myasthenia Gravis (gMG)
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- There're 3 dose groups in this study.Dose will be escalated based on "3+3" rule. (Experimental): There're 3 dose groups in this study for CAR-T cell infusion: 1×10^5/kg, 2×10^5/kg, 3×10^5/kg. Dose will be escalated based on "3+3" rule. 3~6 subjects will be enrolled into each dose group, approximately 9~18 subjects in total will be enrolled. Subjects of each dose group will be observed for DLT within 28 days (Dose-limiting toxicities (DLT) observation period) after GC012F injection infusion.
  Interventions: Drug: GC012F injection

INTERVENTIONS:
Drug: GC012F injection — Subjects will be infused with GC012F Injection within 48-72 hours after lymphodepletion pretreatment, the infusion dose (CAR-T cells) and groups are as follows:
  1. Dose group 1: 1 × 10^5/kg;
  2. Dose group 2: 2 × 10^5/kg;
  3. Dose group 3: 3 × 10^5/kg; Note: For subjects weighing ≤70 kg: number of infused CAR-T cells = (1, 2 or 3) (±20%) × 10^5 × body weight(kg); for subjects weighing >70 kg: number of infused CAR-T cells (fixed doses of GC012F Injection) = (1, 2 or 3) (±20%) × 10^5 × 70 kg.

SUMMARY:
This is a single-arm, open-label and early exploratory clinical study, with the purpose to study the safety, tolerability and initial clinical efficacy of GC012F Injection in the treatment of refractory GMG and to evaluate the PK, PD characteristics and immunogenicity in subjects with refractory GMG infused with GC012F Injection.

DETAILED DESCRIPTION:
This is a single-arm, open-label and early exploratory clinical study, with the purpose to study the safety, tolerability and initial clinical efficacy of GC012F Injection in the treatment of refractory GMG and to evaluate the PK, PD characteristics and immunogenicity in subjects with refractory GMG infused with GC012F Injection.

This study includes periods of screening, apheresis, baseline, lymphodepletion pretreatment, assessment before infusion, infusion of CAR-T cells, and Safety and efficacy follow-ups, long-term follow-ups, and withdrawal of study visits (if any).

Eligible subjects will receive the apheresis and then infusion after the production of CAR-T product. Subjects will receive lymphodepletion pretreatment, and assessments prior to CAR-T cell infusion. Subjects who meet the cell infusion criteria will receive CAR-T cell infusion with the doses specified in the protocol, and the doses in the same group or subsequent group can be adjusted based on the safety and clinical efficacy.

There're 3 dose groups in this study for CAR-T cell infusion: 1×10^5/kg, 2×10^5/kg, 3×10^5/kg. Dose will be escalated based on "3+3" rule. 3~6 subjects will be enrolled into each dose group, approximately 9~18 subjects in total will be enrolled. Subjects of each dose group will be observed for DLT within 28 days (Dose-limiting toxicities (DLT) observation period) after GC012F injection infusion.

After all proposed subjects in each dose group complete the 28-day DLT observation period, the Safety Monitoring Committee (SMC) will evaluate the clinical safety and pharmacokinetic data (if available). Only after obtaining the approval of SMC and collaborator may new subjects be enrolled in the next dose group. Additionally, in order to ensure the safety of CAR-T therapy, the SMC may recommend increasing the frequency of safety committee evaluations according to the safety situation and study progress (e.g., conducting an SMC assessment for each newly enrolled subject).

The dose escalation rules are as follows: Each dose level will enroll 3 to 6 subjects, and only after all subjects in a dose group complete the DLT assessment, meet escalation criteria, and have undergone evaluation by the SMC (considering clinical safety and pharmacokinetic data, if available) and received collaborator approval will they proceed to the next dose level.

The criteria for dose escalation are: if none of the first 3 patients in a group experience DLT during the observation period, the study may proceed to the next dose group. If one patient among the first three experiences DLT during the observation period, three additional patients will be enrolled to the same dose group. If DLT cases are ≤1 out of the total 6 enrolled patients during the DLT observation period, the study can proceed to the next dose group. If the number of DLT cases exceeds 1, dose escalation will be halted (see the table below for details) Number of DLT cases Measures 0/3 Escalation to the next dose group 1/3 Enrolled 3 additional subjects 1/6 Escalation to the next dose group

≥2/3 or ≥2/6 1. Dose escalation will be halted 2. Dose de-escalation to a lower dose level:

1. If only 3 subjects were enrolled at the dose level, 3 additional subjects will be enrolled at that dose level;
2. If there have been 6 subjects at the dose level, DLT cases are ≤1, the dose is MTD.

After all subjects in a dose group have completed the DLT observation period, all clinical study data collected during that period, particularly safety data, will be assessed. Following evaluation and approval by the SMC, which will consider the clinical safety and pharmacokinetic data (if available), the collaborator will decide whether to enroll new subjects in that dose group, halt or continue dose escalation, or introduce an intermediate dose group.

If more than one DLT is observed in the 1×10^5/kg dose group, following approval by the SMC, the researchers and collaborators will discuss whether to explore a lower dose group. If no DLT is observed after escalating to 3×10^5/kg, the decision to explore a higher dose group will be based on a comprehensive review of safety data, CAR-T cell expansion persistence parameters, and efficacy data, after SMC evaluation and approval, followed by discussions between researchers and collaborators.

Given that the activity of cell-based therapies (which are long-lasting) does not show a clear dose dependency, exposure of subjects to excessively low doses may not yield clinical benefit. Therefore, this study will determine or adjust the infusion dose for patients based on the safety of the GC012F injection, parameters for CAR-T cell expansion persistence, and clinical efficacy, following assessment and agreement by the SMC along with further discussions with the researchers and collaborators.

DLT assessments will be performed for evaluable subjects within 28 days post-GC012F injection. Subjects will be replaced if any of the following situations occur during the DLT assessment period: (1) subjects withdraw from the study for reasons not related to DLT, (2) prohibited medications were used prior to DLT occurrence, or (3) safety evaluations required for DLT assessment are not completed.

Following CAR-T cell infusion, subjects will be monitored for safety, cell proliferation persistence, and efficacy, until disease progression, withdrawal from the study with refusal of further follow-up, death, withdrawal of informed consent, loss to follow-up, or 24 weeks post-infusion(whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all the following criteria can be included in this study:

  1. Subjects or their legal representative voluntary signing the ICF, and willing and able to follow the procedure in this study.
  2. Aged between 18 and 75 years old (including 75), no gender limitation;
  3. Patients with confirmed refractory GMG, and the clinical classification according to MGFA is IIa-IVb (including IIa, IIb, IIIa, IIIb, IVa and IVb) at screening;
  4. At screening, the MG-ADL score must be ≥6, with ocular symptoms accounting for less than 50% of the total score, and QMG must be ≥11;
  5. Ineffectiveness of conventional treatment and/or lack of effective therapeutic options, referring to relapse or exacerbation after standard treatments with hormones, immunosuppressants (e.g., azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine A, cyclophosphamide, methotrexate, etc.), or biological agents (e.g., rituximab);
  6. If the subject is currently using corticosteroids, the dose of prednisone must not exceed 30 mg/day (or the equivalent dose of other corticosteroids) and must remain stable for at least 4 weeks prior to infusion;
  7. Only subjects with positive MG-specific autoantibodies: the titer/level of anti-acetylcholine receptor (anti-AChR) antibodies or muscle-specific kinase (anti-MuSK) antibodies must be above the reference laboratory's upper normal limit (UNL);
  8. The results of laboratory test during screening period shall meet all following criteria:

     1. Neu ≥1.0 × 109/L; Hb ≥8.0 g/dL; PLT ≥50 × 109/L;
     2. ALT ≤3 × ULN; AST ≤3 × ULN; TBIL <2 × ULN (DBIL ≤1.5 × ULN for subjects with Gilbert's syndrome)
     3. Creatinine clearance (19.3 Appendix 3) ≥30 mL/min;
     4. APTT ≤1.5 × ULN, PT ≤1.5 × ULN;
     5. LVEF ≥50% based on echocardiography, no findings of pericardial effusion.
  9. Women of childbearing potential (WCBP) should:

     1. Have a negative serum β human chorionic gonadotropin (β-hCG) pregnancy test confirmed by investigators during the screening period;
     2. Agree to avoid breastfeeding during the study period until at least 1 year after the infusion of GC012F Injection or until two consecutive flow cytometry tests show the absence of CAR-T cells (whichever occurs later).
  10. Any male subjects who have sexual partners and female subjects with childbearing potential shall agree to take effective contraceptive methods (e.g. oral contraceptive pills, intrauterine device or condoms) from the screening starting until at least 1 year post GC012F Injection infusion or until two consecutive flow cytometry tests show the absence of CAR-T cells (whichever occurs later). Male subjects must agree to use condoms during sexual contact with pregnant females or females with fertility for at least 1 year after the infusion of GC012F Injection, even if a successful vasectomy has been performed;
  11. Venous access available for blood collection, and no contraindications for leukapheresis.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from the study:

  1. Subjects have a history of severe hypersensitivity or allergy;
  2. Any contraindication for fludarabine, cyclophosphamide and any component of the investigational product;
  3. Administration of intravenous immunoglobulin or plasmapheresis or immunoadsorption treatment within 4 weeks prior to infusion;
  4. Use of B-cell targeting drugs, including but not limited to rituximab, Belimumab, and Telitacicept, within 6 months prior to apheresis;
  5. Used tacrolimus, cyclosporine, azathioprine, mycophenolate, mycophenolate, methotrexate, etc., within 3 weeks prior to apheresis;
  6. Treatment with neonatal Fc receptor (FcRn) antagonists (such as Efgartigimod, etc.) within 3 weeks prior to apheresis
  7. Use of complement inhibition therapy (such as eculizumab, etc.) within 3 weeks prior to apheresis;
  8. Subjects with any of the following heart diseases:

     1. Congestive heart failure (New York Heart Association (NYHA) Class III or IV);
     2. Experienced unstable angina, myocardial infarction or underwent coronary artery bypass grafting (CABG) within 6 months prior to screening period;
     3. Clinically significant ventricular arrhythmias or a history of unexplained syncope not due to vasovagal reaction or dehydration; or a QTc interval >480 ms during screening;
     4. History of severe non-ischemic cardiomyopathy.
     5. Serious cardiovascular abnormalities (such as abnormal brain natriuretic peptide BNP/ troponin and other indicators) and the investigators estimate that the patients should not be enrolled;
  9. Accompanied by other uncontrolled malignant tumors. Subjects with the following conditions will be eligible: early-stage tumors that have received curative treatment (carcinoma in situ or stage I tumors, or non-ulcerated primary melanoma with a depth <1 mm and no involvement of lymph nodes), basal cell skin cancer, skin squamous cell carcinoma, cervical carcinoma in situ, or breast cancer in situ that has received potential curative treatment;
  10. Severe underlying medical conditions, such as:

      1. Fungal, bacterial, viral or other infections or suspected fungal, bacterial, viral or other infections that cannot be controlled or require general intravenous administration (including tuberculosis infection where with clear evidence of disease activity);
      2. Significant clinical evidence of dementia or mental status changes;
      3. History of any central nervous system (CNS) or neurodegenerative diseases, (e.g., epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, psychiatric disorders).
  11. Positive results in any of the following tests:

      1. HIV antibody positive;
      2. HBsAg positive; or HBcAb positive and HBV-DNA above the lower limit of detection of the analytical method;
      3. HCV antibody positive with HCV RNA above the lower limit of detection of the analysis method; or known history of hepatitis C without completion of antiviral therapy for ≥24 weeks;
      4. Syphilis antibody positive.
  12. Received prior therapy of CAR-T for any target;
  13. Previous organ transplant or allogeneic bone marrow transplants;
  14. Surgery within 2 weeks prior to lymphodepletion or planning to have surgery during the study period (except for planned local anesthesia procedures, provided they are not performed within 2 weeks after infusion);
  15. Receipt of a live-attenuated vaccine within 4 weeks prior to lymphodepletion;
  16. Participation in any other clinical trial within 4 weeks prior to signing ICF, or the date of signing the ICF still within 5 half-lives of the drug from the last dose in the last clinical trial (whichever is longer);
  17. Pregnant women or lactating women who do not agree to abstain from breastfeeding, men and women who have a fertility plan during participation in this study or within 1 year after receiving study treatment;
  18. Based on the Columbia-Suicide Severity Rating Scale (C-SSRS), subjects had a current intention to commit suicide, i.e., C-SSRS item 4 on "suicide" (intention to act, But active suicidal ideation without a specific plan) or question 5 (active suicidal ideation with a specific plan and intent) answered "yes" or had a current history of suicidal behavior
  19. Any situation that, in the investigator's judgment, may interfere with the subject's participation in the entire trial, confound trial results, or be contrary to the subject's best interests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2027-02-13 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints | Since signing the ICF until 24-week post-infusion or premature withdrawal from the study, whichever comes first.
  1、DLT incidence;
  DLT is defined as any of the following conditions associated with GC012F Injection occurring within 28 days post cell infusion:
  1. Neurotoxicity: Grade 3 and 4, which cannot recover to Grade 2 or lower within 7 days after therapeutic intervention;
  2. CRS: Grade 4, which cannot recover to Grade 2 or lower within 3 days after therapeutic intervention;
  3. Non-hematological toxicity: Grade 3 and Grade 4, involving heart, lung and kidney, which cannot recover to Grade 2 or lower within 28 days after therapeutic intervention; Grade 5;
  4. Hematological toxicity: Grade 4, which cannot recover to Grade 2 or lower within 3 days after therapeutic intervention. The predictable complication for chemotherapeutics is not included as a DLT in this study.
Primary endpoints | Since signing the ICF until 24-week post-infusion or premature withdrawal from the study, whichever comes first.
  Abnormal results of physical examination, vital signs, laboratory tests, electrocardiography and echocardiography, and the frequency and severity of AEs.
  The grading criteria for adverse event severity were based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0

SECONDARY OUTCOMES:
Secondary endpoints | Since signing the ICF until 24-week post-infusion or premature withdrawal from the study, whichever comes first.
  Disease activity index in 24 weeks after infusion including but not limited to:
  * The improvement and proportion of subjects on MG-ADL score and QMG score from baseline to 24 weeks post-infusion; MG-ADL total score of 24 points. The higher the score, the more serious the impact of the disease on daily life.
  * The improvement and proportion of subjects on MGC from baseline to 24 weeks post-infusion; MGC total score of 50 points. The higher the score, the more serious the impact of the life
  * The mean change of PRO (including MG-QoL15r scores) from baseline to 24 weeks post-infusion; The higher the score, the more serious the impact of the life
  * The change of MGFA post-intervention status from baseline to 24 weeks post infusion;
  * The decrease of titer of pathogenic antibody levels and proportion of subjects from baseline to 24 weeks post-infusion;
Secondary endpoints | Since signing the ICF until Long-term follow-up period or withdraw
  PK parameters of CAR-T cells in peripheral blood (i.e. Cmax, Tmac, AUC, etc.)
  1. GC012F CAR gene copy number in peripheral blood on D-1,D4,D7,D10,D14,D28,D56,D84,D168,D168+84D,D672+84D,OR withdraw
  2. GC012F CAR-T cell count in peripheral blood on D-1,D4,D7,D10,D14,D28,D56,D84,D168,D168+84D,D672+84D,OR withdraw
  3. Anti-GC012F antibody in peripheral blood on D-1,D28,D56,D84,D168,D168+84D,D672+84D,OR withdraw
  4. Lymphocyte subpopulations in peripheral blood and B cell related tests
  5. Tissue or bone marrow (if required) cell cluster related tests
  6. Tissue or bone marrow (if required) CAR-T gene-related tests 4.5.6 are on D-1,D7,D14,D28,D56,D84,D168,D168+84D,D672+84D,OR withdraw
  7. sBCMA in peripheral blood on D-1,D7,D14,D28,D56,D84,D168,D168+84D,D672+84D,OR withdraw
  8. RCL and Lentivirus insertion siteon D-1 M1/3/6/12/18/24, twice a year for 3-5 years and once a year for 6-15 years
Secondary endpoints | Since signing the ICF until 24-week post-infusion or premature withdrawal from the study, whichever comes first.
  Levels of cytokine in peripheral blood [IL-2, IL-6, IL8,IL-10, IL-15, IL-17, IFN-γ, TNF-α, MCP-1and GM-CSF (if applicable), lymphocyte subsets and free BCMA in peripheral blood after GC012F infusion;

OTHER OUTCOMES:
Exploratory endpoints | Baseline to 24 weeks post GC012F infusion;
  The detection rate of CAR-T antibody in peripheral blood from baseline to 24 weeks post GC012F infusion;
Exploratory endpoints | baseline to 24 weeks post GC012F infusion
  The change of patients and serum immunoglobulin concentration (including IgG, IgM, IgA and IgE) from baseline to 24 weeks post GC012F infusion
Exploratory endpoints | on D-1 ,M1/3/6/12/18/24
  Detection rate of RCL.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, affiliated to Fudan University, Shanghai,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Undecided